CLINICAL TRIAL: NCT00318617
Title: A Two Part Study to Separately Evaluate the Effect of 4-week Treatment With GW501516X Relative to Placebo on Cardiac Energetics in a Randomized, Single-blind, Repeat Dose, Parallel Group Design in Healthy Male Subjects
Brief Title: Effect Of GW501516X On How The Heart Obtains And Uses Energy
Status: Terminated | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: PAD100964
Record Dates: First submitted 2006-04-25; First posted 2006-04-27 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Dyslipidaemias; Heart Failure
Keywords: peroxisome proliferator activated receptors,; PPARs,; Heart Failure,; cardiac energetics,; MRI,; GW501516X; fatty acid metabolism,
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Drug: GW510516X

SUMMARY:
The purpose of this study is to determine the effect of a 4-week treatment period with GW501516X on how the heart obtains and uses energy. The energy of the heart will be measured by Magnetic Resonance Imaging (MRI). This study will also measure a number of other potential markers of drug activity, including levels of certain lipids (fats) and proteins in your blood. The data from this study may help researchers better understand the actions of this drug in the body and if this drug may be useful to treat patients with heart disease.

ELIGIBILITY:
Inclusion criteria:

* Non-smoking.
* Body Mass Index of greater than 27 and less than 32 and who weigh 120 kg (264 lbs) or less and have a waist circumference of greater than 95 cm (37.5 inches).

Exclusion criteria:

* History of muscle disease, coagulation disorders, heart disease or abnormal heart rhythm (or a family history of early coronary artery disease).
* Documented diabetes, hypoglycemia, thyroid disfunction or adrenal disorder.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30
Dates: Start 2005-12

PRIMARY OUTCOMES:
Energy-related chemicals and heart contraction, determined by MRI measurement of the heart.

SECONDARY OUTCOMES:
Additional energy-related chemicals, determined by MRI measurement of the heart. Blood proteins. Safety of GW501516X.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Philadelphia, Pennsylvania, United States